CLINICAL TRIAL: NCT04700878
Title: A Randomized Controlled Evaluation of a Compassion-course With the Aim of Reducing Stress of Conscience and Work-related Stress and Increase Levels of Professional Quality of Life and Self-compassion in Healthcare Professionals
Brief Title: A Randomized Controlled Evaluation of a Compassion-course for Healthcare Professionals
Acronym: ICOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Kalmar County Council (Unknown); Sormland County Council, Sweden (Other); Kronoberg County Council (Other Government)
Responsible Party: Principal Investigator, Anna Bratt, PhD, Associate professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-05505
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Psychological Stress; Compassion; Occupational Health; Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The sample size was determined based on an expected between group effect size (between ICOP and ICB) of Cohen's d = 0.4 for the primary outcome at the five-week follow-up for the primary analysis for participants with SCQ scores of 45 and higher. To reach 80% power, the study need 100 participants in each active arm. Expecting 20% attrition, the investigators will include 120 participants. Thirty participants are required in the waitlist group with an expected between-group effect between the ICOP group and the waitlist of d = 0.8. Including the expected attrition, 36 participants will be required. Given the 200 participants and a power of 80%, the non-inferiority analysis will provide a minimal clinically important difference of roughly d = 0.35.
  Participants with SCQ scores below 45 will be included for secondary analyses, thus expect to include 480 participants (ICOP and ICB), with an additional 72 participants in the waitlist group, for a total of 552.
Who Masked: Care Provider
Masking Description: This study is a single-blind randomized trial where eligible participants will informed about that they will be assigned to either of two different stress-management courses or to waitlist, but they are unaware of which particular conditions. The waitlist group (ten weeks waitlist and thereafter either compassion- or cognitive behavioural courses) will receive thorough information about the two different courses and thereafter rate how attractive they find each course. Then they get to choose which course they want to attend to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Internet-based compassion course (Experimental): Therapist guided Internet-compassion course for workrelated stress.
  Interventions: Behavioral: General Internet-based cognitive behavioural course for stress management
- General internet-based CBT stress management course (Active Comparator): Therapist guided Internet-cognitive behavioral (CBT) course for workrelated stress.
  Interventions: Behavioral: General Internet-based cognitive behavioural course for stress management
- Waitlist (Other): Waitlist for 10 weeks, and thereafter the general internet-based CBT management course.
  Interventions: Behavioral: Internet-based compassion course for stress managemant; Behavioral: General Internet-based cognitive behavioural course for stress management

INTERVENTIONS:
Behavioral: Internet-based compassion course for stress managemant — A five week long, structured self-help program with weekly reports to, and feedback from a compassion-focused (CFT) therapist over the Internet. Includes traditional CFT-methods for stress-related problems.
  Arms: Waitlist
Behavioral: General Internet-based cognitive behavioural course for stress management — A five week long, structured self-help program with weekly reports to, and feedback from a cognitive-behavioral (CBT) therapist over the Internet. Includes traditional CBT-methods for stress-related problems.

SUMMARY:
The aim is to investigate whether an internet-based compassion course of five modules contributes to reducing stress of conscience and work-related stress, increase the experience of professional quality of life and self-compassion in healthcare professionals.

DETAILED DESCRIPTION:
Reactions to severe stress is one of the most common causes of sick leave in Sweden. Previous research has shown that compassion interventions for staff can affect work-related stress by increased self-care, better self-awareness and an increased healthy attitude, however, Swedish studies on the subject are scarce.

Compassion is a motivation to reduce suffering in oneself and others characterized by a warm, understanding, and respectful attitude. In addition to beneficial effects for the staff, a compassion-oriented approach, has shown to improve the relationship between patient and staff, increase patient satisfaction with care and reduce patient anxiety and stress. As a result of the covid-19 pandemic, healthcare professionals have been exposed to difficult physical and mental work conditions that cause feelings of stress and inadequacy. In the long run, increased stress can cause fatigue and increased number of sick leaves. This can in turn contribute to increased stress for the staff who remain working and difficulties to recruit new staff, which make the situation worse. There is a lack of interventions for staff aimed at preventing stress-related health issues, enabling recovery and reduce mental suffering linked to a stressful work situations. The aim of this study is to find a method that help healthcare providers cope with stress of conscience in relation to stressful work situations, particularly during the current covid-19 pandemic. A five week internet-based compassion course of five modules will be conducted and evaluated with the aim of exploring whether the course contributes to reduce stress of conscience and work-related stress, and increases the levels of professional quality of life and self-compassion among healthcare professionals. The internet-based compassion course will be compared with: one group that is on a waiting list for ten weeks and then receives an internet-based general stress management course and one group that participate in the general stress management course.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be as follows: the participants work directly with patients full-time or part-time, score 45 points or higher on the primary outcome measure Stress of Conscience Questionnaire (SCQ), are proficient in Swedish, have the requisite time to attend a digital course, and accept the course's format.

The exclusion criteria include being partially or fully on sick leave due to stress.

All criteria are assessed on the basis of self-assessment forms of the participants, but in case of uncertainty, follow-up questions can be done by phone.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change (from baseline) in Stress of conscience | 0, 5, 10 and 15 weeks and 6 months after baseline
  Stress of Conscience Questionnaire (SCQ). The purpose of the SCQ is to estimate stress related to a troubled conscience. The questionnaire consists of nine items describing different healthcare situations, each made up of two parts, an A question and a B question. The A question concerns how frequently the subject estimates that the situation discussed arises in the workplace. This is assessed on a 6-point Likert scale, where 0 is 'Never' and 5 stands for 'Every day'. For each A question, there is a B question following it, in which the degree to which the conscience is troubled in the given situation is estimated on a 10 cm visual analogue scale. The visual analogue scale ranges from 0 = 'No, it gives me no troubled conscience at all' to 5 = 'Yes, it gives me a very troubled conscience'.

SECONDARY OUTCOMES:
Change (from baseline) in Professional quality of life | 0, 5, 10 and 15 weeks and 6 months after baseline
  Professional quality of life scale (PROQOL) Professional quality of life is the quality one feels in relation to their work as a helper. Both the positive and negative aspects of doing one's job influence ones professional quality of life. Professional quality of life incorporates two aspects, the positive (Compassion Satisfaction) and the negative (Compassion Fatigue). Compassion fatigue breaks into two parts. The first part concerns things such like exhaustion, frustration, anger and depression typical of burnout. Secondary Traumatic Stress is a negative feeling driven by fear and work-related trauma. Some trauma at work can be direct (primary) trauma. In other cases, work-related trauma be a combination of both primary and secondary trauma. The PROQOL consists of 30 questions assessed on a 5-point Likert scale, where 0 is 'Never' and 5 stands for 'Very often'.
Change (from baseline) in Work-related stress | 0, 5, 10 and 15 weeks and 6 months after baseline
  Copenhagen Psychosocial Questionnaire (COPSOQ), assessing psychosocial factors at work, stress, and the well-being of employees.
Change (from baseline) in Self-compassion | 0, 5, 10 and 15 weeks and 6 months after baseline
  Self-compassion scale (SCS) consists of 26 items, assessed on a 5-point Likert scale, where 0 is 'Almost never' to 5 for 'Almost always'.

OTHER OUTCOMES:
Sick leave | Number of periods of sick leave according the registry MIDAS from week 5 after baseline until week 52 after baseline.
  Sick leave from MIDAS registry, from the Swedish Social Insurance Agency
Satisfaction with treatment | Week 5 after baseline
  Questions of satisfaction with the internet-based course and treatment credibility scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Bratt, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Linnaeus University, Department of Psychology, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: No